CLINICAL TRIAL: NCT04344730
Title: Dexamethasone and Oxygen Support Strategies in ICU Patients With Covid-19 pneumonia_COVIDICUS
Brief Title: Dexamethasone and Oxygen Support Strategies in ICU Patients With Covid-19 Pneumonia
Acronym: COVIDICUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200388; 2020-001457-43 (EudraCT Number)
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Acute Hypoxemic Respiratory Failure; COVID-19
Keywords: COVID-19; acute hypoxemic respiratory failure (AHRF)
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19 | interventions — Calcium Dobesilate; Respiration, Artificial

STUDY DESIGN:
Intervention Model Description: In non-mechanically ventilated patients, a 2x2 factorial design will be used to assess the two interventions, separately.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking label is available only for the treatment assignation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Standard oxygen 1 (Placebo Comparator): Standard oxygen and placebo of Dexamethasone
  Interventions: Drug: placebo; Procedure: conventional oxygen
- Standard oxygen 2 (Experimental): Standard oxygen and Dexamethasone
  Interventions: Drug: Dexamethasone injection; Procedure: conventional oxygen
- CPAP 1 (Experimental): CPAP and placebo of Dexamethasone
  Interventions: Drug: placebo; Procedure: CPAP
- CPAP 2 (Experimental): CPAP and Dexamethasone
  Interventions: Drug: Dexamethasone injection; Procedure: CPAP
- HFNO 1 (Experimental): HFNO and placebo of Dexamethasone
  Interventions: Drug: placebo; Procedure: HFNO
- HFNO 2 (Experimental): HFNO and Dexamethasone
  Interventions: Drug: Dexamethasone injection; Procedure: HFNO
- mechanically ventilated 1 (Placebo Comparator): placebo
  Interventions: Drug: placebo; Procedure: mechanical ventilation
- mechanically ventilated 2 (Experimental): Dexamethasone
  Interventions: Drug: Dexamethasone injection; Procedure: mechanical ventilation

INTERVENTIONS:
Drug: Dexamethasone injection — Box of 10 DEXAMETHASONE 20 mg / 5 ml, solution for injection in ampoule of 5mL. Each allocated box contains complete treatment from D1 to D10 for one patient.
  Other Names: experimental treatment
  Arms: CPAP 2; HFNO 2; Standard oxygen 2; mechanically ventilated 2
Drug: placebo — Box of 10 NaCl 0,9% , solution for injection in ampoule of 5mL. Each allocated box contains complete treatment from D1 to D10 for one patient.
  Arms: CPAP 1; HFNO 1; Standard oxygen 1; mechanically ventilated 1
Procedure: conventional oxygen — The oxygen flow will be adjusted to maintain an oxygen saturation level of 92% or more, as measured by means of pulse oximetry (SpO2)
  Arms: Standard oxygen 1; Standard oxygen 2
Procedure: CPAP — Patients assigned to the CPAP plus oxygen group will receive periods of CPAP in addition to the standard treatment.The oxygen flow will be adjusted to maintain an oxygen saturation level of 92% or more, as measured by means of pulse oximetry (SpO2)
  Arms: CPAP 1; CPAP 2
Procedure: HFNO — TIn the high-flow-nasal cannula group, oxygen will be delivered through a heated humidifier (Airvo-2, Fisher and Paykel Healthcare) and applied continuously through large-bore binasal prongs, with a gas flow rate of 30 liters per minute and adjusted based on the clinical response. FiO2 will be adjusted for the target SpO2
  Arms: HFNO 1; HFNO 2
Procedure: mechanical ventilation — The oxygen flow will be adjusted to maintain an oxygen saturation level of 92% or more, as measured by means of pulse oximetry (SpO2)
  Arms: mechanically ventilated 1; mechanically ventilated 2

SUMMARY:
The main manifestation of COVID-19 is acute hypoxemic respiratory failure (AHRF). In patients with AHRF, the need for invasive mechanical ventilation is associated with high mortality.

Two hypotheses will be tested in this study. The first hypothesis is the benefit of corticosteroid therapy on severe COVID-19 infection admitted in ICU in terms of survival.

The second hypothesis is that, in the subset of patients free of mechanical ventilation at admission, either Continuous Positive Airway Pressure (CPAP) or High-Flow Nasal Oxygen (HFNO) allows to reduce intubation rate safely during COVID-19 related acute hypoxemic respiratory failure.

DETAILED DESCRIPTION:
The main manifestation of COVID-19 is acute hypoxemic respiratory failure (AHRF). In patients with AHRF, the need for invasive mechanical ventilation is associated with high mortality.

Two hypotheses will be tested in this study. The first hypothesis is the benefit of corticosteroid therapy on severe COVID-19 infection admitted in ICU in terms of survival.

The second hypothesis is that, in the subset of patients free of mechanical ventilation at admission, either Continuous Positive Airway Pressure (CPAP) or High-Flow Nasal Oxygen (HFNO) allows to reduce intubation rate safely during COVID-19 related acute hypoxemic respiratory failure.

The main objective is to assess the impact of dexamethasone on overall mortality at day-60 after randomization in patients admitted in ICU for severe COVID-19 infection.

In non mechanical ventilation (MV) patients, the additional objective is to assess whether oxygen support based on either HFNO or CPAP modality in COVID-19 related AHRF reduces the need for mechanical ventilation at day-28.

An ancillary study CACAO (COVIDICUS air contamination) will be performed in 4 centers aiming at assessing the environmental contamination by SARS-CoV-2 according to the oxygen support modality. Additional funding will be searched for these analyses (submitted for ANR call).

A metanalysis on individual data will be performed using patients enrolled in the 3 PHRC flash exploring the activity of corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admitted to ICU within 48 hours
3. Confirmed or highly suspected COVID-19 infection
4. Acute hypoxemic respiratory failure (PaO2 <70 mmHg or SpO2<90% on room air or tachypnea>30/min or labored breathing or respiratory distress; need for oxygen flow >=6L/min)
5. Any treatment intended to treat the SARS-CoV-2 infection in the absence of contraindications (either as a compassionate use or in the context of a clinical trial, i.e remdesivir, lopinavir/ritonavir, favipiravir, hydroxychloroquine and any other new drug with potential activity).

Non-inclusion Criteria:

1. Moribund status
2. Pregnancy or breastfeeding
3. Long term corticotherapy at a dose of 0.5mg/kg/j or higher
4. Active and untreated bacterial, fungal or parasitic infection
5. Not Written informed consent from the patient or a legal representative if appropriate . If absence a legal representative the patient may be included in emergency procedure
6. hypersensitivity to dexamethasone or to any of the excipients
7. Not Affiliation to the French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The time-to-death from all causes | day-60
  The time-to-death from all causes within the first 60 days after randomization.
The time to need for mechanical ventilation (MV) | day-28.
  the time to need for mechanical ventilation (MV), as defined by any of the 3 criteria for intubation within the first 28 days after randomization.

SECONDARY OUTCOMES:
The viral load in the respiratory tract | day-10
  The cycle threshold for SARS-CoV-2 PCR at baseline, day 7+/-1 and day 10 +/- in samples of the same origin (preferably subglottic i.e. bronchoalveolar lavage or tracheal aspiration, otherwise nasopharyngeal swab)
Number of patient with at least one episode of healthcare-associated infections | day-28
  Proportion of patients with at least one episode of any healthcare-associated infection between randomization and D28
Number of days alive without mechanical ventilation | day-28
  To compare the exposition to mechanical ventilation
Measure of SOFA score | day-1 to day 3, day 7, day 10, day 21, day 28
  Changes in SOFA (Sepsis-related Organ Failure Assessment) score. (min = 0 for normal status max = 24 for worse status)
Number of days alive without renal replacement therapy | day-28
  to compare the exposition to renal replacement therapy
Lengths of ICU-stay | day-60
  To compare the lengths of ICU
Lengths of hospital-stay | day-60
  To compare the lengths of hospital-stay
Number of patients with severe hypoxemia, | day 60
  Proportion of patients with severe hypoxemia, which is defined as an oxygen saturation of less than 80% during the same interval during the interval between induction and 2 minutes after tracheal intubation
Proportion of patients with cardiac arrest within 1 hour after intubation | day 60
  Proportion of patients with cardiac arrest within 1 hour after intubation
Overall survival | day 60
  To compare Overall survival after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jean François TIMSIT, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bichat - Aphp, Paris, France

REFERENCES:
- [Derived] Chevret S, Bouadma L, Dupuis C, Burdet C, Timsit JF; COVIDICUS RCT group. Which severe COVID-19 patients could benefit from high dose dexamethasone? A Bayesian post-hoc reanalysis of the COVIDICUS randomized clinical trial. Ann Intensive Care. 2023 Aug 27;13(1):75. doi: 10.1186/s13613-023-01168-z. PMID 37634234
- [Derived] Chevret S, Timsit JF, Biard L. Challenges of using external data in clinical trials- an illustration in patients with COVID-19. BMC Med Res Methodol. 2022 Dec 15;22(1):321. doi: 10.1186/s12874-022-01769-5. PMID 36522698
- [Derived] Bouadma L, Mekontso-Dessap A, Burdet C, Merdji H, Poissy J, Dupuis C, Guitton C, Schwebel C, Cohen Y, Bruel C, Marzouk M, Geri G, Cerf C, Megarbane B, Garcon P, Kipnis E, Visseaux B, Beldjoudi N, Chevret S, Timsit JF; COVIDICUS Study Group. High-Dose Dexamethasone and Oxygen Support Strategies in Intensive Care Unit Patients With Severe COVID-19 Acute Hypoxemic Respiratory Failure: The COVIDICUS Randomized Clinical Trial. JAMA Intern Med. 2022 Sep 1;182(9):906-916. doi: 10.1001/jamainternmed.2022.2168. PMID 35788622